CLINICAL TRIAL: NCT06924619
Title: A Prospective, Randomized, Controlled Phase Ⅱ Clinical Trial of Neoadjuvant Radiotherapy for Locally Advanced Unresectable Thymoma
Brief Title: Neoadjuvant Radiotherapy for Locally Advanced Unresectable Thymoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Y2024-1244
Record Dates: First submitted 2025-04-06; First posted 2025-04-11 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-01

CONDITIONS: Locally Advanced Thymoma
Keywords: neoadjuvant radiotherapy; Locally Advanced Thymoma; neoadjuvant chemoradiotherapy
MeSH Terms: interventions — Neoadjuvant Therapy; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- the neoadjuvant radiotherapy group (Active Comparator): This group will receive radiotherapy with 40-50 Gy in 20-25 fractions.
  Interventions: Radiation: neoadjuvant radiotherapy
- the neoadjuvant chemoradiotherapy group (Experimental): This group will receive concurrent chemotherapy with radiotherapy. The specific chemotherapy plan is to administer cisplatin intravenously at a dose of 25 mg/m² simultaneously on the first day of radiotherapy, followed by a 6-day rest period. 4-5 cycles of chemotherapy will be conducted, depending on the schedule of the radiotherapy.
  Interventions: Radiation: neoadjuvant radiotherapy; Drug: cisplatin

INTERVENTIONS:
Radiation: neoadjuvant radiotherapy — Target the primary tumor region with 40-50 Gy in 20-25 fractions.
Drug: cisplatin — The cisplatin will be given concurrently with radiotherapy (25 mg/m² , D1, QW) for 4-5 cycles.
  Arms: the neoadjuvant chemoradiotherapy group

SUMMARY:
The goal of this prospective, randomized, controlled phase II clinical study is to evaluate the efficacy and safety of neoadjuvant radiotherapy in patients with locally advanced unresectable thymoma. The main questions it aims to answer are:

1. Which treatment method is more effective in improving the radical resection rate: neoadjuvant chemoradiotherapy or neoadjuvant radiotherapy ?
2. The safety and adverse reactions of neoadjuvant radiotherapy? Does the addition of neoadjuvant chemotherapy have an impact on this?

Participants will be randomly divided into two groups: one group will receive neoadjuvant radiotherapy, and the other will receive neoadjuvant chemoradiotherapy. The primary endpoint of the study is to evaluate the radical resection rate (R0) of two groups. The secondary endpoints will include the pathological complete response rate (pCR), 3-year progression-free survival, and safety and toxicities. In addition, this study will explore the feasibility and completion rate of minimally invasive surgical resection.

DETAILED DESCRIPTION:
For patients with thymoma, surgery is the optimal choice, and it has been proven to improve the survival rate of patients with thymoma. For locally advanced unresectable thymoma, direct surgical resection is associated with significant trauma, a high incidence of surgical complications, and a risk of postoperative recurrence. The application of neoadjuvant therapy is expected to reduce tumor volume and downstage the tumor, thereby increasing the rate of complete tumor resection (R0). Clinical practice has confirmed that thymic tumors are sensitive to both radiotherapy and chemotherapy. However, neoadjuvant chemotherapy regimens for thymoma have not been unified, and the available evidence recommends cisplatin based combination regimens. Earlier retrospective studies mainly targeting locally advanced unresectable thymoma suggested that neoadjuvant radiotherapy could achieve an R0 resection rate of about 50%-75% in these patients. In recent years, neoadjuvant chemoradiotherapy has shown promise in terms of objective response rate and R0 resection rate in patients with thymoma. There is still controversy over how to choose an appropriate neoadjuvant treatment protocol for such patients, and there is a lack of randomized prospective controlled studies.

In this prospective randomized controlled study, participants will be randomly assigned in a 1:1 ratio into two groups. One group will receive neoadjuvant radiotherapy alone, while the other group will receive the same radiotherapy regimen in combination with concurrent cisplatin chemotherapy. Participants in both groups will undergo standard surgery based on efficacy assessment. The purpose of this study is to evaluate the impact of these two approaches on the R0 resection rate in patients and to comprehensively assess the safety of the treatment modalities. This study also aims to provide clinical evidence for neoadjuvant treatment strategies in locally advanced unresectable thymoma.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years and ≤75 years.
* Histologically confirmed thymoma of Masaoka-Koga stage III-IV A.
* Assessed as unresectable thymoma by a thoracic surgeon prior to treatment.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
* No prior anti-thymoma treatment, including but not limited to systemic chemotherapy, radiotherapy, surgery, or immunotherapy.
* Presence of at least one measurable lesion according to RECIST v1.1 criteria.
* Cardiopulmonary function compatible with surgery.
* Expected survival of >3 months.
* Comprehensive evaluation completed within 28 days before enrollment in the study, with a full blood cell test obtained within 15 days, demonstrating normal visceral organ function and normal bone marrow function.
* Negative serum or urine pregnancy test for women of childbearing potential within 14 days before study enrollment.
* Willingness of the patient to sign an informed consent form and to adhere to the specified follow-up schedule.

Exclusion Criteria:

* Histologically confirmed thymic neuroendocrine tumor.
* Currently participating in an interventional clinical study that may affect this study, or having received other investigational drugs or devices within 4 weeks prior to the first treatment in this study.
* Pregnant or breastfeeding women.
* Previous history of thoracic radiotherapy.
* Deemed unsuitable for three-dimensional conformal or intensity-modulated radiotherapy by a radiation oncology specialist.
* History of allogeneic bone marrow or organ transplantation.
* History of malignancies other than thymoma within the past 3 years, or untreated other primary malignancies.
* Serious comorbidities that would affect the study treatment.
* Any history or evidence of disease, treatment, or abnormal laboratory values that could interfere with the study results or prevent the participant from completing the study, or other situations deemed unsuitable for enrollment by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Estimated)
Dates: Start 2024-10-30 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2029-05-01 (Estimated)

PRIMARY OUTCOMES:
Radical resection rate（R0） | up to 1 year
  The tumor lesion is completely resected, with no residual tumor visible to the naked eye at the surgical margins, and no cancer cells detectable at the margins under the microscope.

SECONDARY OUTCOMES:
pCR rate | up to 1 year
  ypT0N0
PFS | up to 3 years
  PFS measures the duration from the initiation of treatment to the point of disease progression, recurrence, or death from any cause.
Safety and toxicities | up to 3 years
  Adverse events will be evaluated according to CTCAE v5.0 .

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang, China